CLINICAL TRIAL: NCT05832541
Title: Expression of Epithelial-Mesenchymal Transition (EMT) Associated Markers in Peri-implant Tissues From Peri-implantitis Patients: A Case-Control Study
Brief Title: Expression of Epithelial-Mesenchymal Transition Associated Markers in Peri-implant Tissues
Status: Recruiting | Type: Observational
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Talib Ali Karam Alnajaty, Principal Investigator, University of Baghdad
Other Study IDs: 535622
Record Dates: First submitted 2023-03-22; First posted 2023-04-27 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Peri-implantitis
Keywords: Peri-implantitis; Peri-implant diseases; Epithelial-mesenchymal transition; E-cadherin; Vimentin
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fixed peri-implant soft tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Test group (peri-implantitis): peri-implant tissue specimen will be taken after identification of diseased interproximal implant sites. Following local anesthesia specimen will be taken either by supracrestal incision to remove all diseased soft tissue surrounding the implant or by making 2 parallel incisions, 4 mm apart, with a 15C scalpel blade through the soft tissue until bone contact would be achieved. The 2 incisions will be connected with a perpendicular incision that will be placed at a distance of 4 mm from the proximal surface of implant. The biopsies, including the entire supracrestal soft tissue portion of the diseased site, will be carefully retrieved and prepared for histopathological and immunohistochemical analysis
- Control group (clinically healthy): tissue sample for control group will be collected from patients undergoing implant surgery. After local anesthesia, a crystal incision will be performed, and a full-thickness flap will be elevated. Following the osteotomy, one or more implants of 4.5-5.0 mm in diameter will be placed. A narrow diameter healing abutment will be screwed in with an insertion torque > 20 NM., and flaps will be repositioned and sutured to obtain optimal adaptation of the mucosa to the titanium abutment.
  Sample harvesting will be done after 2 months of healing using circular punch of 4.5-5.0 mm diameter or performing a circular incision by surgical blade by which a 1.5 mm thick collar of peri-implant soft tissue will be harvested and prepared for histopathological and immunohistochemical analysis. A new 4.5-5.0 mm-wide smooth-surfaced healing abutment will be connected to the implant directly after the biopsy sampling.

SUMMARY:
Peri-implantitis is an inflammation of bacterial etiology characterized by inflammation of mucous membranes and bone loss around the dental implant. A specific dental plaque bacteria could stimulate host cells, including the junctional epithelium, to secrete a range of pro-inflammatory cytokines involved in initiating the epithelial-mesenchymal transition (EMT) process. EMT has been described as the transdifferentiation of epithelial cells into motile mesenchymal cells.

Moreover, cytokines and bacterial products have been highlighted as EMT-predisposing factors. The EMT process could render epithelial cells to lose their cell-cell adhesion and cell polarity that lend these cells to lose their function as an integrated epithelial barrier.

E-cadherin is a calcium-dependent cell adhesion molecule that establishes cell-cell adhesion that plays a critical role in maintaining a barrier function in the human epithelium, including gingiva. The loss of E-cadherin is one of the most common biological indicators for EMT. In contrast, vimentin is an intermediate filament expressed in mesenchymal cells and is a canonical marker for EMT, which also promotes cell motility and an invasive phenotype.

It is largely reported that EMT is regulated by various transcriptional factors such as Snail Family Transcriptional Repressor SNAIL1 and SNAIL2, zinc-finger E-box-binding (ZEB)1 and ZEB2 and TWIST transcription factors that suppress epithelial marker genes, and activate genes related with the mesenchymal phenotype.

Recently, in vivo study has investigated the level of EMT markers in the gingival tissues of periodontitis patients. It was found that the expression of E-cadherin was downregulated while vimentin expression was upregulated.

Despite the similarities and differences between the pathogenesis of periodontal and peri-implant diseases, the role of dental biofilm in the etiopathogenesis of the aforementioned diseases was studied largely. While it is now accepted that EMT may potentially play a role in periodontal disease pathogenicity, the possible role of EMT in the disintegration of the peri-implant epithelial barrier and the pathogenesis of peri-implant disease has not yet been investigated.

DETAILED DESCRIPTION:
Dental implant therapy is a reliable treatment for replacing missing or lost teeth. Despite its high survival and success rates, it has long been realized that biological complications could occur in osseointegrated implants, collectively termed peri-implant diseases. Peri-implantitis is the second most common form of peri-implant disease, and its prevalence was shown to be 10% to 30% at the implant level and 20% at the patient level.

Peri-implantitis is an inflammation of bacterial etiology characterized by inflammation of mucous membranes and bone loss around the dental implant. Clinically, it shows signs of inflammation, bleeding on probing and/or suppuration, increased probing depths, and/or recession of the mucosal margin in addition to radiographic bone loss compared to previous examinations.

Inflammatory peri-implant lesions usually start due to the accumulation of bacterial plaque and progress in a faster pattern compared to periodontitis.

It has been reported that specific dental plaque bacteria could stimulate host cells, including the junctional epithelium, to secrete a range of pro-inflammatory cytokines involved in initiating the epithelial-mesenchymal transition (EMT) process. EMT has been described as the transdifferentiation of epithelial cells into motile mesenchymal cells. It is considered integral in the development, wound healing, and stem cell behavior and contributes pathologically to fibrosis and cancer progression.

Moreover, cytokines and bacterial products have been highlighted as EMT-predisposing factors. It has been proposed that the EMT process could render epithelial cells to lose their cell-cell adhesion and cell polarity that lend these cells to lose their function as an integrated epithelial barrier. Consequently, bacterial invasion into the underlying connective tissues could occur, and epithelial cells are assumed to have a mesenchymal cell phenotype through the upregulation of mesenchymal markers and downregulation of epithelial markers.

E-cadherin is a calcium-dependent cell adhesion molecule that establishes cell-cell adhesion, known as the adherens junction, playing a critical role in maintaining a barrier function in the human epithelium, including gingiva. The loss of E-cadherin is one of the most common biological indicators for EMT. In contrast, vimentin is an intermediate filament expressed in mesenchymal cells and is a canonical marker for EMT, which also promotes cell motility and an invasive phenotype. It has been shown that the level of vimentin protein expression is significantly increased by P. gingivalis infection.

It is largely reported that EMT is regulated by various transcriptional factors such as Snail Family Transcriptional Repressor SNAIL1 and SNAIL2, zinc-finger E-box-binding (ZEB)1 and ZEB2 and TWIST transcription factors that suppress epithelial marker genes, and activate genes related with the mesenchymal phenotype. These transcriptional factors act as E-cadherin repressors and play a pivotal role in development, fibrosis, and cancer. Several signaling pathways collaborate in the beginning and advancement of EMT, and they can promote SNAIL1 expression and transforming growth factor beta.

Recently, in vivo study has investigated the level of EMT markers in the gingival tissues of periodontitis patients. It was found that the expression of E-cadherin was downregulated while vimentin expression was upregulated. Accordingly, the authors proposed that EMT may potentially play an essential role in the pathogenesis and prognosis of periodontal disease.

Much of the etiology and pathogenesis of peri-implant disease was acknowledged to be similar to periodontitis since both share many clinical and radiologic features in common for destructive inflammatory diseases. However, in contrast to periodontitis, peri-implantitis lesions show a poorer vascular supply, a lack of connective tissue encapsulation of large inflammatory cell infiltrates, and a differing cell profile with high numbers of B cells, osteoclasts, and neutrophils. This suggests that peri-implantitis has a similar aetiopathogenesis to periodontitis but also notable differences; its progression seems faster and more aggressive.

Despite these similarities and differences between the pathogenesis of periodontal and peri-implant diseases, the role of dental biofilm in the etiopathogenesis of the aforementioned diseases was studied largely. While it is now accepted that EMT may potentially play a role in periodontal disease pathogenicity, the possible role of EMT in the disintegration of the peri-implant epithelial barrier and the pathogenesis of peri-implant disease has not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

* For test group: adult patient age ≥18 years old presented having at least one dental implant with the following criteria for test group 1: (a) be in function for >12 months; (b) clinically diagnosed as peri-implantitis with probing pocket depth ≥ 6 mm, bleeding on probing and/or suppuration; (c) presence of radiographic bone loss when compared to previous radiographs or with bone loss ≥ 3 mm apical to the 1st thread of the fixture; (d) presence of visual signs of inflammation.
* For the control group: adult patient age ≥18 years old presented with: (a) one or more adjacent missing teeth in the posterior maxilla or mandible (positions premolar to molar); (b) adequate bone quality and availability for an implant placement of 4.5- 5.0 mm diameter and 8.5-13 mm length; (c) keratinized mucosa (KT) width of at least 3 mm.

for both groups the patients give written consent to participate and attend the planned follow-up visits

Exclusion Criteria:

* For the test group: the exclusion criteria will be as follows: (a) patients with a history of chronic diseases such as diabetes mellitus; (b) currently smokers; (c) pregnant or lactating women; (d) patients who received peri-implant surgical therapy within 6 months before sampling; (e) patients who received antimicrobial therapy (systemic or local) within 3 months before sampling.
* For the control group: the exclusion criteria will be as follows: (a) medical condition contraindicating implant surgery; (b) local inflammation (including untreated periodontitis); (c) post-extraction sites with less than 6 weeks of healing; (d) persistent intraoral infection; (e) absence of keratinized tissue; (f) history of chronic diseases such as diabetes mellitus; (g) currently a smoker and former smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants of this study will be selected from the patients' pool who will attend private clinics in Karbala and nearby governorates. The target population will be those who seek dental implant therapy. The control group will involve those who intended for replacing their missing teeth by dental implants. On the other hand, the test group will involve those diagnosed with peri-implantitis and need surgical intervention during follow-up visits
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Peri-implant probing pocket depth (PPD) | Measured at baseline just before performing peri-implant tissue harvesting.
  PPD is the distance (in mm) measured from the Peri-implant mucosal margin to the base of the peri-implant sulcus/ pocket measured by using a periodontal probe, recorded at six sites per implant namely; mesio-facial, mid-facial, disto-facial, mesio-oral, mid-oral and disto-oral.
Radiographic bone level (RBL) | Measured at baseline just before performing peri-implant tissue harvesting.
  RBL is the distance (in mm) measured by periapical digital radiograph using the long-cone parallel technique from the implant platform to the radiographic bone level.
Immunohistochemical expression of EMT-related markers | Measured at baseline
  Immunohistochemical expressions of two EMT-related markers (E-cadherin and vimentin) in peri-implant soft tissue samples collected from patients with peri-implantitis and healthy peri-implant tissue will be measured.

SECONDARY OUTCOMES:
Immunohistochemical expression EMT transcriptional factor | Measured at baseline
  The expression of the EMT transcriptional factor (Snail-1) in peri-implant soft tissue samples collected from patients with peri-implantitis and healthy peri-implant tissue will be measured.
Bleeding on probing (BOP) | Measured at baseline just before performing peri-implant tissue harvesting.
  BOP is measured by inserting a periodontal probe to the bottom of the peri-implant sulcus/ pocket with gentle movement around the implant surface. If bleeding occurs within 30 seconds after probing, the site is given a score (1), and a negative score (0) for the non-bleeding site. BOP is recorded at six sites per implant namely; mesio-facial, mid-facial, disto-facial, mesio-oral, mid-oral, disto-oral.

CONTACTS AND LOCATIONS:
Overall Officials: Talib A Alnajaty, Principal Investigator — University of Baghdad
Locations (1):
- Talib A. Alnajaty, Karbala, Iraq

IPD SHARING:
Plan to Share IPD: Undecided